CLINICAL TRIAL: NCT03947424
Title: Safety and Efficacy of Different Modes of Er:YAG Laser Treatment for Snoring in Comparison With Placebo
Brief Title: Clinical Tial of Er:YAG Laser Snoring Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luis Monteiro (Other)
Responsible Party: Sponsor-Investigator, Luis Monteiro, DMD, Phd, Auxiliar Professor at the IUCS in Periodontal Surgical Clinic, Oral Pathology and Biopathology, Cooperativa de Ensino Superior, Politécnico e Universitário
Organization: Cooperativa de Ensino Superior, Politécnico e Universitário (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16/CE-IUCS/2018
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Snoring
Keywords: laser; Er:YAG; NightLase; Fotona SMOOTH
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Intervention Model Description: Three groups; laser (LP), laser (SMOOTH), control (sham)
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham treatment consists of laser treatment according to the same protocol as active treatment but with no energy applied. Clinical measurements will be performed by an evaluator unaware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1 (Experimental): Long-pulse (LP) Er:YAG laser snoring treatment.
  Interventions: Device: LP Er:YAG
- Experimental 2 (Experimental): Fotona SMOOTH mode Er:YAG laser snoring treatment.
  Interventions: Device: SMOOTH mode Er:YAG
- Control (Sham Comparator): Sham laser snoring treatment with no energy applied.
  Interventions: Device: sham

INTERVENTIONS:
Device: LP Er:YAG — LP Er:YAG applied to oral mucosa
  Other Names: long-pulsed erbium YAG laser; LP NightLase
  Arms: Experimental 1
Device: SMOOTH mode Er:YAG — SMOOTH mode Er:YAG applied to oral mucosa
  Other Names: SMOOTH mode erbium YAG laser; SMOOTH mode NightLase
  Arms: Experimental 2
Device: sham — Er:YAG laser applied to oral mucosa with no energy
  Other Names: placebo
  Arms: Control

SUMMARY:
Two modes of laser (Er:YAG) treatment for snoring will be compared with sham treatment in a randomized clinical trial.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical outcome of snoring treatment using non-ablative Er:YAG laser in comparison with sham laser treatment. Furthermore, to different modes of Er:YAG laser will be compared; a long-pulse mode (LP) and proprietary SMOOTH mode (Fotona, Slovenia).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent form
* Diagnosis of snoring/apnea including partner information
* Age greater than 18 years.
* Apnea-Hypopnea index (AHI) less than 30.
* No significant nasal stenosis.
* Bed partner present

Exclusion Criteria:

* People who refuse to participate in the study
* Presence of concomitant disorders and/or diseases
* Infections in the throat
* current use of photosensitive drugs
* pregnancy
* scarring in the throat
* acute pollen allergies
* epilepsy
* People starting with an extreme diet or weight loss plan
* Patients who do not want to follow post treatment recommendation concerning food and drinks intake
* Larynx obstruction (floppy epiglottis)
* Oropharynx obstruction caused by palatine tonsils (>50%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
NightLase Snoring Questionnaire-Question 1: Snoring severity change from baseline | 6 months
  This questionnaire consists of eight questions, assessing the severity of snoring (the first question) and other problems associated with sleep-disordered breathing (questions 2-8). Answers will be graded on 11-point scales (0-10) .

SECONDARY OUTCOMES:
Change from baseline in snoring value | 1 month
  Snorelab software used to record snoring
Change from baseline in snoring value | 3 months
  Snorelab software used to record snoring
Change from baseline in snoring value | 12 months
  Snorelab software used to record snoring
Change from baseline in snoring value | 6 months
  Snorelab software used to record snoring
NightLase Snoring Questionnaire-Question 1: Snoring severity change from baseline | 3 months
  This questionnaire consists of eight questions, assessing the severity of snoring (the first question) and other problems associated with sleep-disordered breathing (questions 2-8). Answers will be graded on 11-point scales (0-10) .
NightLase Snoring Questionnaire-Question 1: Snoring severity change from baseline | 12 months
  This questionnaire consists of eight questions, assessing the severity of snoring (the first question) and other problems associated with sleep-disordered breathing (questions 2-8). Answers will be graded on 11-point scales (0-10) .
NightLase Snoring Questionnaire-Question 1: Snoring severity change from baseline | 1 month
  This questionnaire consists of eight questions, assessing the severity of snoring (the first question) and other problems associated with sleep-disordered breathing (questions 2-8). Answers will be graded on 11-point scales (0-10) .
NightLase Snoring Questionnaire change from baseline | 1 month
  This questionnaire consists of eight questions, assessing the severity of snoring (the first question) and other problems associated with sleep-disordered breathing (questions 2-8). Answers will be graded on 11-point scales (0-10) .
NightLase Snoring Questionnaire change from baseline | 3 months
  This questionnaire consists of eight questions, assessing the severity of snoring (the first question) and other problems associated with sleep-disordered breathing (questions 2-8). Answers will be graded on 11-point scales (0-10) .
NightLase Snoring Questionnaire change from baseline | 6 months
  This questionnaire consists of eight questions, assessing the severity of snoring (the first question) and other problems associated with sleep-disordered breathing (questions 2-8). Answers will be graded on 11-point scales (0-10) .
NightLase Snoring Questionnaire change from baseline | 12 months
  This questionnaire consists of eight questions, assessing the severity of snoring (the first question) and other problems associated with sleep-disordered breathing (questions 2-8). Answers will be graded on 11-point scales (0-10) .
Change in EpWorth somnolence scale from baseline | 1 month
  The level of daytime sleepiness in the patients was assessed using the 24-point Epworth scale. Values 0-10 are considered normal, and values 11-24 represent increasing levels of 'excessive daytime sleepiness'.
Change in EpWorth somnolence scale from baseline | 3 months
  The level of daytime sleepiness in the patients was assessed using the 24-point Epworth scale. Values 0-10 are considered normal, and values 11-24 represent increasing levels of 'excessive daytime sleepiness'.
Change in EpWorth somnolence scale from baseline | 6 months
  The level of daytime sleepiness in the patients was assessed using the 24-point Epworth scale. Values 0-10 are considered normal, and values 11-24 represent increasing levels of 'excessive daytime sleepiness'.
Change in EpWorth somnolence scale from baseline | 12 months
  The level of daytime sleepiness in the patients was assessed using the 24-point Epworth scale. Values 0-10 are considered normal, and values 11-24 represent increasing levels of 'excessive daytime sleepiness'.
Change in Quality of life Questionnaire score from baseline | 1 month
  Oral Health Impact Profile-14 on the scale from 0 to 56 with higher scores indicating a poorer oral health-related quality of life.
Change in Quality of life Questionnaire score from baseline | 3 months
  Oral Health Impact Profile-14 on the scale from 0 to 56 with higher scores indicating a poorer oral health-related quality of life.
Change in Quality of life Questionnaire score from baseline | 6 months
  Oral Health Impact Profile-14 on the scale from 0 to 56 with higher scores indicating a poorer oral health-related quality of life.
Change in Quality of life Questionnaire score from baseline | 12 months
  Oral Health Impact Profile-14 on the scale from 0 to 56 with higher scores indicating a poorer oral health-related quality of life.
Change in Apnea - Hypopnea Index (AHI) from baseline. | 3 months
  Measured by polysomnography.
Change in O2 saturation (%) from baseline. | 3 months
  Measured by polysomnography.
Change in snoring time (mean duration of episode in s) from baseline. | 3 months
  Measured by polysomnography.
Change in percentage snoring time of total sleep time (%) from baseline. | 3 months
  Measured by polysomnography.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Monteiro, DMD, PhD, Principal Investigator — Instituto Universitário de Ciências da Saude, CESPU
Locations (1):
- Instituto Universitário de Ciências da Saude, CESPU, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No